CLINICAL TRIAL: NCT00342069
Title: Facilitating Informed for Prenatal Testing: The Role of Ambivalence
Brief Title: Prevalence of Ambivalence Regarding Prenatal Testing
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905067; 05-HG-N067
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Pregnancy
Keywords: Decision Making; Genetic Counseling; Pregnancy Options; Attitudes Toward Reproductive Options; Beliefs About Down Syndrome Risk; Down Syndrome Risk; Pregnancy

SUMMARY:
This study will examine how women think and feel about prenatal testing (amniocentesis and chorionic villus sampling), how those thoughts and feelings change over time, and how they contribute to the decision whether or not to undergo prenatal testing.

Prenatal diagnostic testing is offered to pregnant women at increased risk of carrying a baby affected with a genetic or chromosomal abnormality. Although these tests are well established, standard-of-care procedures, much remains unknown about how best to ensure that women make decisions about whether or not to undergo testing that are consistent with their beliefs and values. This study will explore the extent to which women are ambivalent about prenatal testing and determine how they might benefit from counseling aimed at improving the quality of their decision-making.

Women 18 years of age and older who are scheduled for a prenatal genetics visit at clinics in Baltimore, MD; Minneapolis, MN; Binghamton, NY; Salt Lake City, UT; Washington, DC; and Bellevue, WA, and are at increased risk for having a baby with trisomy 21 (Down syndrome) may be eligible for this study.

Participants complete two short questionnaires and a telephone interview about their thoughts and feelings regarding prenatal testing. The first two surveys examine the women's thoughts and feelings before and after prenatal counseling. Both are completed at the prenatal clinic-one before and one after the counseling session. The third survey is done by telephone a few weeks after the prenatal visit to find out if the participant did or did not have prenatal testing and learn about her thoughts and feelings regarding her decision.

DETAILED DESCRIPTION:
The proposed study seeks to estimate the prevalence of ambivalence about undergoing diagnostic testing among women referred for prenatal genetic counseling, and the predictors and decisional consequences of such ambivalence. Women seen at six different U.S. prenatal clinics for genetic counseling at increased risk for carrying a fetus with trisomy 21 [N=240] will be asked to complete a questionnaire on three occasions: prior to counseling; immediately after counseling, and later by telephone. These data will be used to describe the extent to which a sample of U.S. women referred for prenatal counseling based upon maternal age or results of a screening test are ambivalent about prenatal testing and might benefit from interventions aimed at improving the quality of decision-making.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women must be equal to or greater than or equal to 18 years of age, speak English and be competent to consent to participate in the study.

Participants must be pregnant women at increased risk for carrying a fetus with trisomy 21 determined by maternal age or an abnormal screening test, such as ultrasound and/or triple tests.

EXCLUSION CRITERIA:

Women will be excluded form participation if they have ever previously undergone prenatal (in current pregnancy or in a past pregnancy) or participated in prenatal genetic counseling.

Women will also be excluded from the study if they have a family history (at least one first degree relative) of a genetic condition and are seeking prenatal testing for genetic indication including trisomy 21.

Women at increased risk for other chromosomal or genetic conditions will be excluded.

Children and men are excluded as women are the patients in prenatal genetics clinic and the ultimate decision-makers about prenatal testing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12-17; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Georgetown University, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Genetic Counsel Program, Binghamton, New York
  - University of Utah, Salt Lake City, Utah
  - Eastside Maternal Fetal Medicine, Bellevue, Washington

REFERENCES:
- [Background] Conner M, Povey R, Sparks P, James R, Shepherd R. Moderating role of attitudinal ambivalence within the theory of planned behaviour. Br J Soc Psychol. 2003 Mar;42(Pt 1):75-94. doi: 10.1348/014466603763276135. PMID 12713757